CLINICAL TRIAL: NCT01637129
Title: Transcranial Magnetic Stimulation in Children With Stroke
Acronym: TMSCS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Warren Lo, Associate Clinical Professor of Pediatrics and Neurology, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB11-00324; 273611 (Other Grant/Funding Number: RINCH)
Record Dates: First submitted 2012-06-25; First posted 2012-07-10 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Hemiparesis; Neonatal Stroke; Ischemic Stroke; Hemorrhagic Stroke; Thrombotic Stroke
Keywords: Childhood stroke; Perinatal stroke; Pediatric stroke; Presumed perinatal stroke; Children who have hemiparesis
MeSH Terms: conditions — Paresis; Ischemic Stroke; Hemorrhagic Stroke; Thrombotic Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic Stimulation (Active Comparator): Active Magnetic Stimulation with repetitive transcranial magnetic stimulation
  Interventions: Device: Transcranial Magnetic Stimulation
- No Intervention (Placebo Comparator): Sham Magnetic Stimulation
  Interventions: Device: Sham Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation, repetitive at 1Hz
  Other Names: MagStim
  Arms: Magnetic Stimulation
Device: Sham Magnetic Stimulation — Sham Magnetic Stimulation
  Other Names: MagStim
  Arms: No Intervention

SUMMARY:
This is a pilot study of repetitive transcranial magnetic stimulation (rTMS) to test tolerance and efficacy in children who have hemiparesis from acquired or presumed perinatal stroke.

DETAILED DESCRIPTION:
The investigators will begin to test the hypothesis that rTMS will be tolerated and will result in improved hand strength and mobility when compared with sham stimulation.

Aim 1: To determine whether 1 Hz rTMS applied to the hemisphere opposite the infarct (contralesional or healthy hemisphere) is tolerated by children ages 6-18 years who have chronic motor sequelae from a stroke.

Aim 2: To determine whether 8 sessions of inhibitory 1 Hz rTMS to the contralesional healthy hemisphere improves grip strength and hand mobility when compared with sham stimulation in controls.

ELIGIBILITY:
Inclusion Criteria:

1. A history of ischemic or hemorrhagic stroke at least 6 months prior to recruitment, and causing current unilateral motor impairment of hand function (scoring 1-3 on a modified Ashworth scale; scale explained in Appendix).
2. Cerebral infarction spares the transcallosal pathways.
3. Cerebral injury confirmed by brain MRI or CT
4. Ages 6-18 years inclusive.

Exclusion Criteria:

1. The presence of an implanted device such as a pacemaker, vagal nerve stimulator, or recently implanted cardiovascular stent; arterial aneurysms; arteriovenous malformations; obstructive hydrocephalus.
2. Infarction of the cortical motor areas.
3. Presence of a brain tumor or suspected neurodegenerative disease.
4. Intractable epilepsy or a history of poorly controlled epilepsy.
5. Current use of medications that may lower seizure threshold (such as specific antipsychotics, specific antidepressants, amphetamines)
6. Hand function limited to rigid flexion or extension (score = 4 on the modified Ashworth scale)
7. Disorders causing hallucinations, delusions, or excessive anxiety or depression.
8. Pre-existing chronic pain syndromes including intractable headache and chronic daily headache.
9. Pregnancy.
10. Any sensorimotor or cognitive impairment that prevents valid responses on study measures.
11. Bilateral strokes (cerebral injuries) involving motor cortex and/or corpus callosum
12. All patients and parents must be naïve regarding the effects and sensations of rTMS (i.e., patients and/or parents with prior exposure to TMS will be excluded).
13. Subject has had a recent neurosurgical procedure involving the brain.
14. Subject suffered traumatic brain injury that places the subject at risk of seizures.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Tolerance to repetitive stimulation | Up to 2 days
  The patient's reports of side effects recorded on the CRF at each session will be tabulated and the pre-stimulation scores will be subtracted from the post-stimulation scores.
  Cognitive function will be assessed with 6 measures (Executive Function / Spatial Problem Solving, Psychomotor Function / Speed of Processing, Visual Attention / Vigilance, Visual Learning & Memory, Verbal Learning & Memory, and Attention / Working Memory measures). As with the tolerance assessments, we will tabulate before-stimulation and after-stimulation assessments and analyze the difference.

SECONDARY OUTCOMES:
Upper extremity strength and mobility | Up to 2 Months
  Upper extremity strength will be assessed with a Jtech dynamometer at three different locations: elbow extension (triceps), elbow flexion (biceps), and grip.
  Joint mobility at the elbow and wrist will be assessed with the modified Ashworth score.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Lo, MD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University School of Health and Rehabilitation Sciences, Columbus, Ohio